CLINICAL TRIAL: NCT01892982
Title: Improving Preterm Outcomes by Safeguarding Maternal Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Tufts Medical Center (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-31407; R01HD072069 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Depression; Child Development
Keywords: Maternal Depression; Preterm Birth; Preterm Outcomes; Child Development
MeSH Terms: conditions — Depression; Premature Birth

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem Solving Education tailored to NICU (Experimental): NICU-PSE integrates motivational interviewing and problem solving, with ongoing monitoring and linkage to mental health services for mothers with worsening depressive symptoms over time. The intervention is provided over six sessions, including three tailored, post-discharge sessions, which address issues common to families of preterm infants: caregiver burden, complexity of medical follow-up, and social reintegration following hospitalization.
  Interventions: Behavioral: Problem Solving Education tailored to NICU
- Control (No Intervention): Both study groups receive standard NICU medical, social work, and nursing services. At each study site, attending neonatologists and pediatrics residents constitute the medical team, and all families are assigned a social worker.

INTERVENTIONS:
Behavioral: Problem Solving Education tailored to NICU
  Arms: Problem Solving Education tailored to NICU

SUMMARY:
The investigators' goal is to optimize the developmental outcomes of preterm infants by preventing depression and improving functioning among their mothers during the critical first year of life. The investigators are conducting a randomized controlled trial of a replicable, lay-delivered intervention - the basic approach of which is to use an empirically-supported, cognitive behavioral strategy to help mothers solve their unique daily problems and address some of the predictable challenges to parenting a preterm infant.

DETAILED DESCRIPTION:
Preterm infants are born at biological risk for poor health and developmental outcomes; and those born to low-income families face additional social risks known to further interfere with healthy child development. In its 2006 report, Preterm Birth, the Institute of Medicine (IOM) stated the public health importance of optimizing the developmental outcomes of preterm infants, and specifically called for novel postnatal intervention strategies to accomplish this goal. Our proposed strategy is based on the premise that preventing maternal depression - and optimizing maternal functioning in specific domains that mediate the relationship between maternal depression and adverse child effects - will ultimately improve the developmental outcomes of this vulnerable child population.

Problem Solving Education (PSE) is a cognitive behavioral strategy that aims to impart recipients with skills to reduce the impact of stress on personal functioning, and thereby prevent depression. The present project is a randomized trial of a 6-session intervention based on PSE. the investigators aim to enroll 325 mother-infant dyads in four NICUs - Boston Medical Center, Tufts Medical Center, Beth Israel Deaconess Medical Center, and Brigham and Womens Hospital. Over 12-months of follow-up, the investigators will assess the effects of PSE on a series of outcome measures for mothers, a series of measures that represent risk mechanisms by which maternal depression is theorized to impact young children, and a series of child functioning measures.

1. Primary aims. Regarding outcomes for mothers, the investigators aim to:

   1. Decrease the incidence of major depressive episode (MDE) and improve depressive symptom trajectories during the first postpartum year; and
   2. Improve general and parental functioning, as measured by valid and reliable scales.
2. Secondary aims. Regarding risk mechanisms and child outcomes, the investigators aim to:

   1. Improve mothers' sense of mastery, and decrease their caregiver burden and social isolation;
   2. Improve adherence to evidence-based quality indicators for NICU follow-up care;
   3. Improve maternal sensitivity and mother-child interaction patterns; and
   4. Improve infant social engagement, emotionality, and cognitive functioning.
3. Exploratory aims. the investigators will explore the role of a brief set of potential intervention moderators:

   1. On the infant level: severity of infant illness.
   2. On the maternal and family level: maternal trauma history, extended family functioning, and intervention adherence.

ELIGIBILITY:
Inclusion Criteria:

* Baby is 26-34 weeks gestational age
* Baby qualifies to receive Medicaid
* Mother comfortable in English or Spanish
* Singleton or twin gestation
* Baby is expected to survive

Exclusion Criteria:

* Mother in major depressive episode or endorses suicidality
* Mother with psychosis or otherwise cognitively limited
* Mother with known active substance use; custody of infant uncertain
* Infant is critically ill
* Triplets or higher number gestation
* Mother who is enrolled in another study receiving the same intervention that we are testing

Max Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 325 (Actual)
Dates: Start 2013-06; Primary Completion 2018-05-25 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of major depressive episode and depressive symptom trajectories | one year
  To measure depression and depressive symptom trajectories, we will combine a dimensional measure (the Quick Inventory of Depressive Symptoms - QIDS) with the diagnostic Structured Clinical Interview for DSM-IV Disorders (SCID). Administering the QIDS every other month during this time frame will allow us to follow depression symptom trajectories with a repeated measure sensitive to change with treatment. Administering the SCID at 12-months will allow us to determine timing and severity of major depressive episode(s).
General Functioning | one year
  General functioning will be measured by the mean total SAS-SR score, and mean scores for the family, partner, and social SAS subscales. The SAS will be administered at 6 and 12 months of follow-up.

SECONDARY OUTCOMES:
Caregiver burden, mastery and social support | one year
  The Coping Health Inventory for Parents is a valid and reliable instrument designed to measure parents' response to managing family life when they have an ill child. It will be administered together with the Pearlin Mastery Scale and the Medical Outcomes Survey Social Support Scale. Administration of these scales will occur at 6 and 12 months of follow-up.
Adherence to recommended NICU follow-up care | one year
  We assess the following measures of adherence to NICU follow-up care:
  * timing and receipt of health supervision visits and immunizations following NICU discharge - including Palivizumab (Synagis).
  * ratio of complaint-based to preventive primary care visits; evaluation for, and attendance to, early intervention services.
Parent-child interaction | one year
  We will videotape and microcode a 10-minute mother-infant free play session according to the parent, infant, and dyadic scales of the Coding Interactive Behavior Manual (CIB). We will assess the following composites: maternal sensitivity; intrusive and withdrawn maternal interactions; and depressed mood and positive affect.
Socio-emotional functioning | one year
  We will assess the CIB infant social engagement composite. We will assess negative infant emotionality using the 4-minute 'Mask Task' of the Laboratory Temperamental Assessment Battery (Lab-TAB).
Cognitive functioning | one year
  We will use the MacArthur-Bates Communicative Development Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverstein, MD, MPH, Principal Investigator — Boston Medical Center
Locations (4):
- United States (4):
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elansary M, Zuckerman B, Patts G, Antonio J, Mayes LC, Silverstein M. Posttraumatic Stress Symptoms and the Quality of Maternal-Child Interactions in Mothers of Preterm Infants. J Dev Behav Pediatr. 2022 Dec 1;43(9):e605-e613. doi: 10.1097/DBP.0000000000001122. Epub 2022 Aug 29. PMID 36040801